CLINICAL TRIAL: NCT05476471
Title: The Short Effectiveness of Self-Management Skills and Health Promotion Programs on the Health Status of the Pre-frail Individuals in the Communities
Brief Title: The Effectiveness of Health Promotion Programs on the Pre-frail Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shu-Hung Chang (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor-Investigator, Shu-Hung Chang, Professor, Chang Gung University of Science and Technology
Organization: Chang Gung University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZRRPF3J0031
Record Dates: First submitted 2022-07-22; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Older Adults
Keywords: multicomponent exercise training; older adults; physical activity; physical performance; Pre-frailty; Coronavirus Disease 2019 pandemic
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The intervention consisted of one 60-minutes group exercise session once a week in first 8 weeks, and self-management in next 8 weeks. The control arm received an education leaflet.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention arm (Experimental): The intervention consisted of one 60-minutes group exercise session once a week in first 8 weeks, and self-management in next 8 weeks
  Interventions: Behavioral: multicomponent exercise training program
- control arm (No Intervention): The control arm received an education leaflet.

INTERVENTIONS:
Behavioral: multicomponent exercise training program — One supervised 60 minutes training sessions per week were organized combining warm-up, speed-walking, resistance exercise, static and dynamic balance. Supervised walking sessions were for 10-20 minutes at a target intensity of 13-15 on the Borg scale. Thereafter, 10 resistance exercises targeting lower body, trunk and upper body muscles were performed with elastic band. In addition, participants were instructed to accumulate 150 minutes per week of moderate intensity aerobic activity in bouts of at least 10 minutes, and at least 2-3 days all major muscle groups training.
  Arms: intervention arm

SUMMARY:
This pilot study aimed to examine the efficacy of a home-based multicomponent exercise training program in older community- dwellers during to the Coronavirus Disease 2019.

DETAILED DESCRIPTION:
This pilot study aimed to examine the efficacy of a home-based multicomponent exercise training program in older community- dwellers during to the Coronavirus Disease 2019.

Design: A two-arm parallel cluster randomized controlled trial. Older adults ≥60 years old were recruited from eight community units in northern Taiwan. One-hundred and sixty-seven eligible subjects consented to participate in the study. Community units were randomly assigned to either an intervention arm (n=82) or a control arm (n=87). The intervention consisted of one 60-minutes group exercise session once a week in first 8 weeks, and self-management in next 8 weeks. The control arm received an education leaflet. Assessments were performed at baseline and 16 weeks for physical activity, physical performance, and pre-frailty rate. Analysis of covariance or chi-square test adjusted for pretest evaluated the differences between the two study arms.

ELIGIBILITY:
Inclusion Criteria:

* older adult with age ≥ 60 years
* community-dwelling
* no hearing and visual acuity difficulties

Exclusion Criteria:

* Unconscious
* Cognitive impairment or dementia

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Physical activity | 4 month follow up
  International Physical Activity Questionnaire (IPAQ)
short physical performance battery | 4 month follow up
  sit-to-stand, standing balance, and gait-speed
Frailty | 4 month follow up
  Frailty measurement used study of osteoporotic fracture index (SOF)

SECONDARY OUTCOMES:
upper limb muscle strength | 4 month follow up
  hand-grip strength
static balance ability | 4 month follow up
  single-leg standing with the eyes open
physical agility and dynamic balance ability | 4 month follow up
  Timed-Up and Go and Functional Reach Test

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Hung Chang, Ph. D, Principal Investigator — Chang Gung University of Science and Technology
Locations (1):
- Taoyuan, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang SH, Chiang CC, Chien NH. Efficacy of a multicomponent exercise training program intervention in community-dwelling older adults during the COVID-19 pandemic: A cluster randomized controlled trial. Geriatr Nurs. 2023 Jan-Feb;49:148-156. doi: 10.1016/j.gerinurse.2022.11.019. Epub 2022 Dec 16. PMID 36528997